CLINICAL TRIAL: NCT03909399
Title: Prevention and Prophylaxis (Thromboprophylaxis - ACT) of Cancer Associated Thrombosis (CAT) in High Risk Oncology Patients: ACT4CAT.
Brief Title: Prevention and Prophylaxis of Cancer Associated Thrombosis in High Risk Oncology Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hellenic Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: ACT4CAT
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-07

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Vena Cava Thrombosis; Iliac; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevention and Prophylaxis (Thromboprophylaxis - ACT) of Cancer Associated Thrombosis (CAT) in High Risk Oncology Patients: ACT4CAT.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), which includes both deep venous thrombosis (DVT) and pulmonary embolism (PE), is a highly prevalent complication of malignancy. The development of VTE in cancer patients is associated with several adverse consequences including worsened short- and long-term prognosis and survival, mortality, morbidity, chemotherapy postponement, potential hospitalization, need for long-term anticoagulation with attendant bleeding complications and high rates of recurrent VTE . In addition, VTE leads to significant consumption of health care resources; in one study of cancer patients, the adjusted mean incremental all-cause health care costs of VTE were $30,538 per patient. Therefore, the optimal prevention and treatment of VTE are crucial components of patient care in this population. Currently, Low-Molecular-Weight Heparin (LMWH), is the gold standard for the CAT management for the last 15 years Moreover, in a variety of high-risk thrombosis clinical settings, LMWHs agents are safe and effective in preventing VTE. Multiple randomized trials of thromboprophylaxis have been conducted focusing on ambulatory cancer patients receiving chemotherapy. ESMO and ASCO current guidelines suggest considering thromboprophylaxis in high-risk ambulatory cancer patients with LMWHs. ECOG index, metastatic malignancy, chemotherapy and history of thrombosis were significantly associated with the decision to use thromboprophylaxis in most situations.

Additionally, in 2016 Hellenic Society of Medical Oncology (HeSMO) has conducted the GMaT study to assess the awareness of Thrombosis and highlight the current clinical practice in Greece. The study has precluded adoption of outpatient prophylaxis in largely unselected patients with cancer without significant adverse events. Based on GMaT findings, the investigators will proceed in an observational study focusing on thromboprophylaxis in cancer patients with high thrombotic cancer types. In particular, the title of this new study will be "Prevention and Prophylaxis (Thromboprophylaxis - ACT) of Cancer Associated Thrombosis (CAT) in High Risk Oncology Patients: ACT4CAT".

ELIGIBILITY:
Inclusion criteria

* Patients who were diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic, genitourinary or CNS).
* Patients who have already started on thromboprophylaxis treatment according to the current clinical practice guidelines and the clinical judgment of treating physician after discussion with patient, within three months before the study enrollment.
* Age ≥ 18 years
* ECOG 0-2
* Life expectancy >6 months
* Signed informed consent

Exclusion criteria

* Patients who were not diagnosed with histological confirmed high thrombotic risk cancers (GI, thoracic, gynecologic, genitourinary or CNS).
* Patients who have not already started on thromboprophylaxis treatment according to the current clinical practice guidelines or who have already started on thromboprophylaxis but more than three months before the study enrollment.
* Age < 18 years
* ECOG >2
* Life expectancy <6 months
* Not signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The objective of the "ACT4CAT" study is to collect real world data of daily clinical practice regarding thromboprophylaxis in high thrombotic risk ambulatory cancer patients. In particular, in this study we will collect data from patients with high thrombotic risk solid tumors (GI, thoracic, gynecologic, genitourinary or CNS) who receive or not anticancer treatment and have already administered thromboprophylaxis treatment according to the current clinical practice guidelines. Based on these real world data we will try to assess the efficacy and safety of long term VTE thromboprophylaxis in cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Recording all objectively confirmed VTE events for 500 patients during the treatment period | 1 YEAR
  Recording the rate of symptomatic distal deep vein thrombosis (DVT), symptomatic or incidental proximal DVT (including iliac and vena cava thrombosis), symptomatic or incidental pulmonary embolism (PE) or both DVT and P, will also be recorded the agent, the dose and the duration of the antithrombotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Society of Medical Oncology, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided